CLINICAL TRIAL: NCT00431223
Title: Does Computerized Cognitive Skills Training Change Brain Activation Patterns in Schizophrenia?
Brief Title: Brain Activation Patterns in Schizophrenia After Computerized Cognitive Skills Training
Acronym: fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Clinical Director, Manhattan Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05I/C52
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia
Keywords: fMRI; working memory; schizophrenia; treatment refractory; cognitive skills training; dorsolateral prefrontal cortex; cognitive remediation; treatment refractory schizophrenia of > 5 years duration
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Group (Active Comparator): 7 patients were assigned to Cognitive Remediation Therapy..
  Interventions: Behavioral: Cognitive remediation therapy
- Control Group (No Intervention): 4 patients were assigned to Control group or no cognitive remediation therapy.

INTERVENTIONS:
Behavioral: Cognitive remediation therapy — 36 sessions of computerized cognitive skills training over a 12 week duration. 7 patients were assigned to cognitive remediation therapy or CRT Group.
  Other Names: CRT Group
  Arms: Active Group

SUMMARY:
This project is a novel exploratory research project to investigate changes in activation patterns of the dorsolateral prefrontal cortex (DLPFC) in inpatients with schizophrenia who received a 12-week computerized cognitive remediation (CRT) program. The hypothesis is that patients receiving CRT will show greater increase in activation patterns in the brain as compared to controls, and the degree of brain activation will correlate with improvements in working memory.

DETAILED DESCRIPTION:
Abnormalities in the domains of attention, working memory (WM) and information processing are important features of schizophrenia. There is growing literature that cognitive remediation therapy (CRT) can produce modest improvements in cognitive functioning in schizophrenia, suggesting that systematic efforts at improving cognitive functioning are feasible. Cognitive improvement after CRT may correlate with changes in brain activation patterns in specific areas.

After screening, patients are randomized to a 12 week trial of CRT using COGPACK (Marker Software), or to a 12-week control condition. All patients attend 3 weekly 1-hour laboratory sessions, with 1 discussion session per week.

Patients continue their antipsychotic treatment with a typical or atypical antipsychotic during the CRT and 4 weeks prior to enrollment in the study (Phase A). Following Phase A they receive baseline evaluations, including an cognitive activation task (N-back visual-letter task) while being scanned for fMRI , MATRICS neuropsychological test battery, and psychiatric, social functioning, and symptoms assessment.

Patients then enter Phase B with randomization to control or CRT for 12 weeks (36 laboratory sessions). Upon successful completion of 36 sessions, endpoint evaluations include an N-back task while fMRI scan, MATRICS, psychiatric, and social functional assessments.

All baseline and endpoint fMRI scans are conducted at the Center for Advanced Brain Imaging (CABI) at Nathan Kline Institute for Psychiatric Research.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient status
* Age 18 - 55
* Male gender (females are enrolled but will not be scanned)
* DSM-IV diagnosis of schizophrenia (all subtypes) and schizoaffective disorder
* illness duration > 5 years
* MMSE score > 24 (inclusive) at screening
* Stable dose of oral atypical antipsychotic for at least 4 weeks prior to study entry
* Total PANSS score > 60 at screening
* Capacity and willingness to give written informed consent
* Patients deemed not ready to be discharged within the next 12 weeks

Exclusion Criteria:

* Inability to read or speak English
* Documented disease of the central nervous system
* History of intellectual impairment pre-dating onset of symptoms of psychosis (e.g. mental retardation)
* Clinically significant or unstable cardiovascular, renal, hepatic, gastrointestinal, pulmonary, or hematological conditions; HIV positive
* Any medical condition rendering the subject unable to receive an fMRI scan

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Brain activation changes after stimulation with a neurocognitive task in the dorso-lateral prefrontal cortex (DLPFC) | 12 weeks

SECONDARY OUTCOMES:
Examine the relationship of changes in DLPFC activation patterns in relation to improvement on neurocognitive tests | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Kaushik, MD, Principal Investigator — Manhattan Psychaitric Center; Jean-Pierre Lindenmayer, MD, Study Chair — Manhattan Psychiatric Center; Susan McGurk, PhD, Study Chair — Dartmouth College, Hanover; Craig A. Branch, PhD, Study Chair — Center for Advanced Brain Imaging, NKI
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

REFERENCES:
- [Background] Wykes T, Reeder C, Corner J, Williams C, Everitt B. The effects of neurocognitive remediation on executive processing in patients with schizophrenia. Schizophr Bull. 1999;25(2):291-307. doi: 10.1093/oxfordjournals.schbul.a033379. PMID 10416732
- See also: FMRIB Software Library — http://www.fmrib.ox.ac.uk/fsl/
- See also: Wikipedia entry for fMRI — http://en.wikipedia.org/wiki/Functional_magnetic_resonance_imaging